CLINICAL TRIAL: NCT03441828
Title: Effects of Depth of Neuromuscular Block on Surgical Operating Conditions and on Time to Discharge From Post-anesthesia Care Unit in Patients Undergoing Gynecologic Laparoscopic Surgery: a Randomized Prospective Clinical Trial
Brief Title: Effects of Depth of Neuromuscular Block on Surgical Operating Conditions in Gynecologic Laparoscopic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Edoardo De Robertis, Associate Professor, Federico II University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Registro MISP n.54876
Record Dates: First submitted 2018-02-07; First posted 2018-02-22 (Actual); Last update posted 2020-12-04 (Actual); Status verified 2020-12

CONDITIONS: Neuromuscular Blockade

STUDY DESIGN:
Intervention Model Description: After enrollment, patients will be randomized in the two study groups:
  Deep Neuromuscular Block group (group DNMB) Moderate Neuromuscular Block group (group MNMB)
Who Masked: Care Provider
Masking Description: in the assessment of the surgical field quality surgeons are blind respect the level of neuromuscular block received by patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group DNMB (Experimental): Deep Neuromuscular Block group Intervention: maintenance of a deep neuromuscular block by infusion of rocuronium at the starting dose of 0.3-0.6 mg / kg / h, titrated to maintain a TOF count of 0, and a PTC between 1-2.
  Quality of surgical field conditions' assessed by a blind surgeon as a 5 points scale (Optimal= 5 points/ Good= 4 points / Adequate= 3 points / Poor = 2 points / Inadequate = 1 point)
  Interventions: Procedure: Quality of surgical field conditions; Drug: Deep Neuromuscular Block
- Group MNMB (Active Comparator): Moderate Neuromuscular Block group Intervention: maintenance of a moderate neuromuscular block. neuromuscular blockade will be maintained with intravenous bolus of rocuronium (0.15-0.25 mg/kg) titrated to obtain a TOF count of 1-3.
  Quality of surgical field conditions' assessed by a blind surgeon as a 5 points scale (Optimal= 5 points/ Good= 4 points / Adequate= 3 points / Poor = 2 points / Inadequate = 1 point)
  Interventions: Procedure: Quality of surgical field conditions; Drug: Moderate Neuromuscular Block

INTERVENTIONS:
Procedure: Quality of surgical field conditions — evaluation of the intraoperative surgical conditions assessed by the surgeon as a 5 points scale (Optimal= 5 points/ Good= 4 points / Adequate= 3 points / Poor = 2 points / Inadequate = 1 point) given by deep vs moderate neuromuscular block
  Other Names: surgical field
Drug: Deep Neuromuscular Block — maintenance of a deep neuromuscular block by infusion of rocuronium
  Other Names: deep relaxation
  Arms: Group DNMB
Drug: Moderate Neuromuscular Block — maintenance of a moderate neuromuscular block.
  Other Names: moderate relaxation
  Arms: Group MNMB

SUMMARY:
Comparison of the impact of a deep neuromuscular blockade (TOF count = 0 and posttetanic count [PTC] 1-2) and a moderate neuromuscular blockade (TOF count= 1 - 3) on intraoperative surgical conditions assessed by the surgeon as a 5 points scale (Optimal= 5 points/ Good= 4 points / Adequate= 3 points / Poor = 2 points / Inadequate = 1 point) in patients undergoing laparosopy for benign gynecological pathologies.

DETAILED DESCRIPTION:
Objectives.

The primary outcome of the study is to compare the impact of a deep neuromuscular blockade (TOF count = 0 and posttetanic count [PTC] 1-2) and a moderate neuromuscular blockade (TOF count= 1 - 3) on intraoperative surgical conditions assessed by the surgeon as a 5 points scale (Optimal= 5 points/ Good= 4 points / Adequate= 3 points / Poor = 2 points / Inadequate = 1 point).

The use of low intraabdominal pressure (IAP) and its impact on the surgical operating conditions has not yet been adequately defined in the literature, although, it is reasonable to consider that a deep neuromuscular blockade may be beneficial1, especially in gynecologic laparoscopic surgery.2, 3

Secondary outcome is to compare the time to discharge from post-anesthesia care unit (PACU) assessed with the WAKE© score.4 As per protocol adopted in our institution, patients are evaluated with the Modified Aldrete Score5 before discharging from PACU. However the WAKE© score , whichis constructed from the basic 10-point Modified Aldrete Score, addsthe "Zero Tolerance Criteria". In fact, the WAKE© score assigns a score from 0 to 2 to motor function, blood pressure, level of consciousness, respiratory function and oxygen saturation (with a maximum score of 10), plus the Zero Tolerance Criteria which address the presence or absence of pain, postoperative nausea and vomiting (PONV), shivering, pruritus, and orthostatic symptoms. A patient can be discharged from PACU when the WAKE© score is ≥ 9 and when there are not present any zero tolerance criteria (no pain, PONV, shivering, pruritus, and orthostatic symptoms).

The use of low IAP associated with the use of a deep neuromuscular blockade may improve the respiratory function and reduce the postoperative pain and PONV,1, 6-8 thus reducing the time spent in PACU.

Clinical hypotheses.

The use of deep neuromuscular blockade may improve the surgical operating conditions and reduce the time spent in PACU by applying a lower intraabdominal pressure. Sugammadex may be useful to rapid reverse the neuromuscular block. Therefore, discharge time may be reduced. Even if all the surgical procedures in this study will be performed as inpatient surgery, some of this may be possibly performed as outpatient surgery. Evaluating the time to discharge may be relevant, especially for ambulatory surgery, as the cost may be reduced when the time spent in PACU is reduced.9

Laparoscopic surgery requires the formation of the surgical field within the peritoneal cavity by insufflating CO2, and creating a pneumoperitoneum. This type of procedure is not free of adverse effects10 related to insufflation of CO2 and IAP that can induce changes in liver function, hemodynamic and respiratory compromise.11, 12 Moreover, the use low pneumoperitoneum pressure (<12 mmHg) is associated with a significant reduction of postoperative pain.13 The optimization of the surgical field during laparascopic surgery can be achieved with a deep neuromuscular block, using low pressure of insufflation.1 The benefit of using a deep neuromuscular blockade to improve the conditions of laparoscopic surgery is still controversial.14

This study is a single center, prospective clinical trial. Patients scheduled for gynecologic laparoscopy surgery with planned duration less than 60 min, will receive a deep (TOF count = 0 and posttetanic count -PTC- 1-2) or a moderate neuromuscular blockade (TOF count= 1 - 3) according to clinical routine. 50 patients will be studied

Inclusion criteria will be:

* Patients who give written informed consent to the study
* Age: 18-60 years
* ASA risk class: I - II
* Elective gynecologic laparoscopic surgery lasting <60 min (excision of ovarian cyst, endometriosis)

Exclusion criteria will be:

* Lack of consent
* Body Mass Index (BMI)> 30 Kg/m2
* Patients with renal and hepatic dysfunction
* Neuromuscular disorders
* Known hypersensitivity to study drugs
* Pregnant patients
* Conversion to laparotomy

All patients will be hospitalized (inpatient surgery). One hour before surgery, all the subjects included in the study will receive 75 mg diclofenac SC, whilst ranitidine 100 mg IV and ondansetron 4 mg IV will be administered as premedication before entering in the operating room. Standard monitoring will be applied before induction of anesthesia: ECG, pulse oximetry, non-invasive blood pressure, BIS, acceleromyography at the adductor pollicis muscle (TOF-Watch SX ®). A balanced general anesthesia will be adopted. Propofol 2mg/kg and fentanyl 4mcg/kg IV will be administered during induction.

After calibration and stabilization of the TOF-Watch, tracheal intubation will be facilitated with rocuronium bromide 1.2 mg/kg in the DNMB, and 0.6 mg/kg in the MNMB. Anesthesia will be maintained with inhalation of a mixture of air / oxygen 50%/50%, and sevoflurane titrated to obtain a BIS value between 40 - 60. Neuromuscular block will be maintained intraoperatively by a) a continuous intravenous infusion of rocuronium at the starting dose of 0.3-0.6 mg / kg / h , titrated to maintain a TOF count of 0, and a PTC between 1-2; b) neuromuscular blockade will be maintained with intravenous bolus of rocuronium (0.15-0.25 mg/kg) titrated to obtain a TOF count of 1-3. PTC will be evaluated every 5 min, whilst TOF every 15 sec.

After insertion of the Veress needle, pneuomoperitoneum will be accomplished with a set pressure up to 15 mmHg, but reduced to a value of 9 mmHg after all trocar placements. After every 15 min from pneumoperitoneum and at the end of the procedure (before desufflation of pneumoperitoneum), surgeon will be asked to judge the surgical conditions with a five points scale (Optimal= 5 points/ Good= 4 points / Adequate= 3 points / Poor = 2 points / Inadequate = 1 point). In case of inadequate or poor surgical field that hampers surgery, pneumoperitoneum pressure will be increased to 12 mmHg and a bolus of rocuronium will be given as judged appropriate by the attending anesthesiologist. In this case, the final score (which is the average of all values) will be automatically 1 (inadequate). At the end of surgery, after careful desufflation of pneumoperitoneum, sugammadex 4mg/kg in DNMB or 2mg/kg in MNMB will be administered, and patients will be extubated when TOF-ratio >0.9. In PACU, the WAKE© score will be evaluated every 5 mins. When the score is ≥ 9 and the zero tolerance criteria (pain, PONV, shivering, pruritus, and orthostatic symptoms) are not present, patients will be discharged to ward.

For postoperative pain, diclofenac 50 mg SC will be given after 12 hours from the last administration with paracetamol 1 gr IV q 6h starting at the end of surgery. Tramadol 1mg/kg IV will be given as a rescue therapy.

The study will necessitate at least 1 year from IRB approval.

Variables/Time Points of Interest Primary outcome is the evaluation of the intraoperative surgical conditions assessed by the surgeon as a 5 points scale (Optimal= 5 points/ Good= 4 points / Adequate= 3 points / Poor = 2 points / Inadequate = 1 point).

Every 15 min from pneumoperitoneum and at the end of the procedure, surgeon will be asked to judge the surgical conditions with this five points scale.

Secondary outcome is to compare the time to discharge from PACU assessed with the WAKE© score. The WAKE© score will be assessed every 5 minutes from the arrival of the patient in PACU.

Statistical Methods The data analysis will be based on the intent-to-treat approach. The primary end-point of the study is the influence of the depth of the NMB on the surgical conditions assessed by a 5 points scale. For each patient, the final score will be the average of all values (assessed every 15 min from pneuomoperitonuem and at the end of surgery). The analysis on the final score will be tested using a t-test or a Wilcoxon-Mann-Whitney test, using R version 2.15.2 (R: A Language and Environment for Statistical Computing, Vienna, Austria), with a P-value<0.05 considered significant. Data will be presented as mean (SD) or median (IQR), as judged appropriate.

The secondary end-point evaluates the difference in time spent in PACU between the two groups. The analysis will compare the average times to reach a WAKE© score ≥ 9 plus the absence of the "zero tolerance criteria" (pain, PONV, shivering, pruritus, and orthostatic symptoms) of the two groups. The WAKE© score will be assessed every 5 minutes from the arrival of the patient in PACU. The analysis will be tested using a t-test or a Wilcoxon-Mann-Whitney test, using R version 2.15.2 (R: A Language and Environment for Statistical Computing, Vienna, Austria), with a P-value<0.05 considered significant. Data will be presented as mean (SD) or median (IQR), as judged appropriate.

Power/Sample Size:

Based on previous studies,13, 15 a sample size of 50 patients would allow us to detect a clinically relevant difference in the proportion of optimal surgical space conditions during the entire procedure with a power of 80% and a type 1 error risk (α) of 5%.

ELIGIBILITY:
Inclusion Criteria:

* Patients who give written informed consent to the study
* Age: 18-60 years
* ASA risk class: I - II
* Elective gynecologic laparoscopic surgery lasting <60 min (excision of ovarian cyst, endometriosis)

Exclusion Criteria:

* Lack of consent
* Body Mass Index (BMI)> 30 Kg/m2
* Patients with renal and hepatic dysfunction
* Neuromuscular disorders
* Known hypersensitivity to study drugs
* Pregnant patients
* Conversion to laparotomy

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
impact of a deep neuromuscular blockade on surgical conditions | during surgery
  impact of a deep neuromuscular blockade (TOF count = 0 and posttetanic count [PTC] 1-2) and a moderate neuromuscular blockade (TOF count= 1 - 3) on intraoperative surgical conditions assessed by the surgeon as a 5 points scale

SECONDARY OUTCOMES:
the time to discharge from post-anesthesia care unit | first 12 h post op
  the time to discharge from post-anesthesia care unit (PACU) assessed with the WAKE© score (WAKE Score "0-10". Criteria: Blood Pressure / Heart Rate 2 - 1 - 0 ; Movement 2 - 1 - 0; Mental Status 2 - 1 - 0; Respiratory 2 - 1 - 0; O2 Saturation 2 - 1 - 0)

CONTACTS AND LOCATIONS:
Overall Officials: Edoardo De Robertis, PhD, Prof, Principal Investigator — University Federico II
Locations (1):
- University Federico II - AOU, Napoli, Italy

IPD SHARING:
Plan to Share IPD: No
individual participant data will be stored locally

REFERENCES:
- [Derived] Coviello A, Ianniello M, Buonanno P, Di Falco N, Iacovazzo C, Maresca A, Vargas M, Marra A, Candice A, Saccone G, Zullo F, Servillo G. Effects of depth of neuromuscular block on surgical operating conditions in women undergoing gynecologic laparoscopic surgery: a randomized clinical trial. J Anesth Analg Crit Care. 2023 Jan 19;3(1):2. doi: 10.1186/s44158-023-00086-7. PMID 37386582